CLINICAL TRIAL: NCT06060288
Title: Diagnostic Accuracy of Mobile Phone Imaging Compared to Conventional Clinical Examination for Oral Cancer Screening
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mary Fayez Farag Mikhail, Resident Doctor in Department of Oral Medicine ,diagnosis and Periodontology , Faculty of Dentistry Fayoum University, Cairo University
Other Study IDs: 14081996
Record Dates: First submitted 2023-09-23; First posted 2023-09-29 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Premalignant Lesion; Oral Cancer
Keywords: teledentistry; oral cancer screening; oral potentially malignant lesions
MeSH Terms: conditions — Mouth Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Diagnosis by mobile phone imaging — The photographs will be taken with a smartphone iPhone 14 Pro in a one-year period. Imaging will follow the recommendations regarding intraoral photography in oral mucosal screening set by (Lin et al., 2021).
  Personal data and a brief description of the present illness concerning the main complaint will be informed by the patients and recorded in a diagnosis chart of the Oral medicine department Cairo University. Complete intraoral physical examination will be performed by the main investigator under supervision of the main supervisor and the co-supervisor using dental equipment with artificial light.
  Other Names: smartphone iPhone 14 Pro

SUMMARY:
The aim of study is to evaluate the sensitivity and specificity of using mobile phone photographs versus conventional clinical examination as a screening tool for early detection of oral cancer.

DETAILED DESCRIPTION:
Tele-dentistry is a method of providing oral healthcare and dental services through real-time transmission of clinical information using electronic medical records, digital imaging, photography, ICT, and the internet. Oral medicine is a dental specialty that uses tele-dentistry services to manage patients with systemic diseases and comorbidities. However, some oral disorders may have systemic consequences, necessitating additional diagnostic techniques and skilled doctors. Issues such as lack of oral medicine specialists, inexperienced community health workers, and inadequate training for managing complex oral conditions also pose challenges. Delayed diagnosis of oral cancers in underserved communities, poor patient management, high transportation costs, and lengthy waiting lists are some of the challenges faced by patients.

The COVID-19 pandemic has further complicated these issues, causing disruptions in educational programs and access to oral medicine services. Tele-dentistry can facilitate efficient communication between patients and healthcare professionals for various purposes. There is limited research on using tele-dentistry in oral medicine, especially for results like accuracy. Consequently, the present study is designed to evaluate the sensitivity and specificity of using mobile phone images versus conventional clinical examination as a screening tool for early detection of oral cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients have any visible oral mucosal lesions including:

  1. Normal Variants
  2. Reactive and inflammatory lesions
  3. Potentially malignant lesions (PML)
  4. Oral cancer

Exclusion Criteria:

- 1. Patients unable to open their mouth properly due to trismus, pain, fibrosis or scleroderma.

2. Patients unable to follow instructions such as mental disability and children below 12-year-old.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: - Patients have any visible oral mucosal lesions including normal variants, reactive and inflammatory lesions and potentially malignant lesions (PML)
Sampling Method: Non-Probability Sample
Enrollment: 174 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Categorization of oral mucosal lesions | one year
  to categorize the oral lesions into:
  1. Normal variance
  2. Reactive or inflammatory lesions
  3. Potentially malignant lesions
  4. Oral cancer

SECONDARY OUTCOMES:
Referral decision | one year
  when to take a decision of referral to a specialist

CONTACTS AND LOCATIONS:
Overall Officials: Mary F Mikhail, TA, Principal Investigator — master candidate in Cairo University

IPD SHARING:
Plan to Share IPD: Undecided
Data will be available upon request

REFERENCES:
- [Background] Haron N, Zain RB, Nabillah WM, Saleh A, Kallarakkal TG, Ramanathan A, Sinon SH, Razak IA, Cheong SC. Mobile Phone Imaging in Low Resource Settings for Early Detection of Oral Cancer and Concordance with Clinical Oral Examination. Telemed J E Health. 2017 Mar;23(3):192-199. doi: 10.1089/tmj.2016.0128. Epub 2016 Aug 19. PMID 27541205
- [Background] Lin I, Datta M, Laronde DM, Rosin MP, Chan B. Intraoral Photography Recommendations for Remote Risk Assessment and Monitoring of Oral Mucosal Lesions. Int Dent J. 2021 Oct;71(5):384-389. doi: 10.1016/j.identj.2020.12.020. Epub 2021 Feb 20. PMID 33618833